CLINICAL TRIAL: NCT05005481
Title: Incidence and Factors Affecting the Development and Outcome of Phantom Limb Pain (PLP) - A Single-centre Prospective Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Diana Chan Xin Hui (Unknown); Lin Xufeng (Unknown); Yap Haoyun (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021/2456
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NIL intervention — NIL intervention will be performed on patients.

SUMMARY:
Phantom limb pain (PLP), defined as pain felt in the missing portion of the amputated limb following amputation, occurs in a significant percentage of patients who undergo limb amputation and it is among the most difficult chronic pain syndromes to treat. Its incidence has been reported to be around 70% though a local pilot study in 2013 reported the incidence to be 25%. The investigators aim to determine the actual incidence of PLP by conducting a single-centre prospective cohort study and identify risk factors associated with PLP. Subsequently, the investigators will use identified risk factors to develop and validate a risk prediction model for PLP after amputation surgery and design interventional studies aimed at reducing the development of PLP in high risk patients.

DETAILED DESCRIPTION:
Specific aims:

By using prospective design and validated multidimensional pain questionnaire, the investigators aim to better estimate the true incidence of PLP, other associated risk factors and the severity of functional impairment.

This study is divided into 2 phases, of which the first phase of the study would be covered by the scope of the grant.

Phase 1 Primary Aim 1. To determine the local incidence of PLP at 3 months post amputation surgery (as literature suggests that PLP is most likely to develop within 3 months of amputation surgery) Hypothesis It is hypothesized that the incidence of PLP is estimated to be 41-85% from the literature .

Secondary Aims 1. Analyse and delineate modifiable and non-modifiable risk factors (patient, anaesthetic and surgical factors) contributing to the development of PLP. 2. Identify factors likely to prevent or reduce the development of PLP after amputation surgery 3. To identify factors prognosticating patient outcomes and recovery from PLP.

Phase 2 (out of the scope of the grant) Aims:

1. To follow up patients prospectively to identify the long-term functional and psychological effects of PLP on patients

Background information:

According to International Association for the Study of Pain (IASP), Phantom limb pain (PLP) is defined as pain felt in the absent body part. PLP occurs in a significant percentage of patients who undergo limb amputation and it is among the most difficult chronic pain condition to treat. Undertreated PLP, together with other persistent chronic pain secondary to amputation can lead to limitations in both physical and psychosocial function and impair their rehabilitation.

The true prevalence of PLP among people with amputation is unclear, especially among Asian population. There are various reports of PLP prevalence ranging from 40% to 80% depending on the site of amputation, the patient population, and the time since amputation.

The exact reason why some patients develop phantom pain after amputation is still unknown. The development of PLP is likely multifactorial and includes peripheral, central, and psychological factors. Several risk factors associated with the development of PLP have been identified in various studies but the overall results are rather conflicting. Risk factors such as persisting pre-operative pain, stump pain, patient comorbidity contribute to the onset of PLP. The majority of these studies, however, are based on Caucasian population.

Nevertheless, it is increasingly clear that patients with PLP will continue to rise locally in view of higher prevalence of Diabetes Mellitus and malignancy, largely attributed to ageing population. In Singapore, major lower extremity amputation rate has increased from 11.0 per 100,000 population in 2008 to 13.3 per 100,000 population in 2013. It was reported in 2001 that approximately 700 lower extremity amputation (LEA) were performed in patients with diabetes annually. The figures more than doubled to 1500 LEA annually in 2017, due to complications arising from diabetes.

Despite anticipating PLP to be a significant burgeoning healthcare burden, PLP is underreported and undertreated, leading to poor rehabilitation outcome. There is also a paucity on local data, with only one ever publication related to PLP in Singapore. The lack of local data in terms of definitive incidence estimate in our population, the functional impairment from PLP and potential risk factors has greatly hindered the development or implementation of effective interventions for preventing or treating PLP. Thus, the primary aim of this study is to establish the incidence of PLP in our local population, the risk factors associated with PLP and its functional impact.

ELIGIBILITY:
Inclusion criteria for recruitment of patients:

* Age 21-80 years old
* Provided consent for the study
* Types of amputation surgery included: Forefoot amputation, below knee amputation, above knee amputation

Exclusion criteria:

* Cognitive impairment/ uncommunicative patients
* Existing psychiatric condition

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients listed for limb amputation surgery will be recruited in the ward
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Phantom Limb Pain | 3 months
  Phantom Limb Pain

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other institution